CLINICAL TRIAL: NCT02631148
Title: Effects of Melatonin Supplementation on Renal Physiology in a Habitual Sleep Restricted Population.
Acronym: MAST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: International shortage of the chemical para-aminohippuric acid (PAH) due to manufacturing changes, led to inability to perform key measurements to meet trial objectives
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ciaran McMullan, Instructor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015P002161
Record Dates: First submitted 2015-11-13; First posted 2015-12-16 (Estimated); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Prediabetic State
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Melatonin (Experimental): Circadin, controlled release melatonin tablet 2mg by mouth each day before bedtime for 6 weeks
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo tablet identical to Circadin by mouth each day before bedtime for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 2mg controlled release melatonin tablet
  Other Names: Circadin
  Arms: Melatonin
Drug: Placebo — placebo tablet identical to circadin
  Arms: Placebo

SUMMARY:
In a 6 week pilot study, 20 individuals with habitual sleep restriction will all be asked to extend their nightly sleep by 1 hour, and will then be randomized 1:1 to nightly controlled-release oral melatonin (2mg) or placebo. The investigators will assess whether sleep extension and nightly melatonin supplementation in the community is a feasible intervention with a beneficial effect on the following chronic kidney disease (CKD) risk factors: systemic and renal specific renin-aldosterone-angiotensin system (RAAS) activation (systemic plasma renin activity, plasma angiotensin II levels, 24-hour urine aldosterone excretion, and renal plasma flow response to captopril); nocturnal blood pressure measured by 24-hour ambulatory blood pressure monitor; central blood pressure measured by pulse wave analysis; and glucose metabolism measured by Minimal Model assessment of insulin resistance and β-cell response to a mixed meal protocol.

DETAILED DESCRIPTION:
The investigators will recruit individuals from the Boston area who meet the inclusion and exclusion criteria. The investigators will include both men and women and all races and ethnicities. The only exception will be women who are pregnant because certain medications used during the inpatient evaluations (e.g., nitroglycerine), and certain study medications (i.e., captopril) are contraindicated during pregnancy.

Participant Enrollment

Responders to advertisements will be pre-screened by telephone to obtain a body mass index (BMI) estimate and a medical history to gauge potential eligibility. For participants who may be eligible following this phone query, the basic study schema will be described to identify those who remain interested in participation after learning the duration, inpatient requirements, and potential medication use. These individuals will then be invited to attend an outpatient screening visit.

The pilot study is a double-blind, placebo-controlled randomized trial, in which 16 subjects with obesity (body mass index [BMI] ≥30 kg/m2), pre-diabetes (hemoglobin A1C [HbA1C], 5.7-6.4%), and self-reported short sleep duration (<7 hours/night) are randomly assigned 1:1 to receive either placebo or 2 mg of controlled-release melatonin, taken orally every evening 1 hour before bed for 6 weeks. All subjects will be asked to extend their sleep time by one hour during the 6 week period between inpatient visits. Endpoints will be measured at both the baseline and 6-week inpatient visits.

Screening Visit: Screening visits will take place at the Brigham and Women's Outpatient Center for Clinical Investigation During the outpatient screen, Dr. McMullan will explain the study in detail, review the consent form, and answer questions. After obtaining written informed consent for participation, a history and physical examination will be performed in order to initially judge eligibility based upon the criteria set out in that section of this record. Participants deemed potentially eligible based upon the screening history and exam will undergo phlebotomy and analysis for HbA1c, serum chemistries and glucose, and complete blood count (CBC) to confirm eligibility using the criteria presented in the table.

Study Procedures Pre-admission: All participants will wear a wrist activity monitor for a total of 8 weeks; 2 weeks prior to the baseline inpatient visit and for the 6 weeks between inpatient visits. Participants will complete a daily sleep log during the 2 weeks preceding each visit. Three days before admission, participants will be placed on a high salt diet by supplementing their usual diet with 150 millimoles (mmol) sodium/day for 3 days using dry bouillon added to food.

Treatment assignments: Prior to admission for the baseline visit, participants will be randomized (1:1) to receive study medication (melatonin 2mg of controlled release formulation or placebo). All participants will be asked to extend their sleep time by one hour during the 6 week period between inpatient visits.

Baseline and Follow-up inpatient visit: Baseline and 6-week inpatient visits will be virtually identical. Each inpatient visit will begin at 4:00PM on Day 0 and end at 4:00 PM on Day 1.

Day 0 - All participants will begin 24 hour urine collection on admission to the Brigham and Women's Hospital Center for Clinical Investigation (CCI) on the evening of day 0. The 24-hour urine collection will be continued overnight (nurses will keep the daytime (8AM to 8PM) and nighttime (8PM to 8AM) urine separate to permit analysis of diurnal variation in urinary analytes). Subjects will fast after 9 pm to ensure a 12-hour fast by the next morning.

Day 1 -At 8 am, central blood pressure and vascular compliance will be assessed, followed at approximately 9 am by measurement of renal specific RAAS activity via para-aminohippurate (PAH) renal plasma flow testing with captopril, and systemic renin-aldosterone-angiotensin system (RAAS) will be measured by plasma renin activity (PRA), plasma angiotensin II (Ang II) and urine aldosterone. Next the participant will receive a mixed meal (10kcal/kg, 45% carbohydrate, 15% protein, 40% fat, 1g/kg glucose) to be consumed in 15 minutes with blood draws at 0, 10, 20, 30, 60, 90 and 120 minutes from the time the meal had begun to be consumed. Plasma glucose, insulin and c-peptide will be measured in all 7 samples of blood. The 24-hour urine collection will conclude at 4 pm on day 1 and will be used to measure 24-hour excretion of sodium and aldosterone. Finally the participant will be fitted with a Spacelabs 90207 ambulatory blood pressure (BP) monitor prior to discharge to be worn for 24-hours.

Follow-up - During the study, participants will be phoned weekly by a study coordinator to assess for compliance and potential side effects. Dr McMullan will call all subjects every 2 weeks to discuss difficulties encountered with their new sleep schedule, to recommend improvements and encourage compliance with the protocol.

Parameters Measured: At the inpatient visits, the following measurements will be made:

Renal Specific renin-aldosterone-angiotensin system (RAAS) - The activity of the local kidney RAAS can be measured by examining the change in effective renal plasma flow (RPF) after oral captopril while in high sodium balance. Effective RPF is measured as clearance of para-aminohippuric acid (PAH), because PAH is cleared solely and nearly entirely by the kidney. The protocol to measure PAH clearance is performed with the participant supine.

Systemic renin-aldosterone-angiotensin system (RAAS) - plasma renin activity (PRA) and angiotensin II (Ang II) levels will be measured on the first morning blood draw.

Central Blood Pressure - Will be measured using pulse wave analysis using the SphygmoCor system (AtCor Medical, West Ryde, New South Wales, Australia), which measures central blood pressure and arterial stiffness.

Glucose metabolism - Will be evaluated by applying the Oral Minimal Model method to the results of a 2 hour 7- measurement, mixed meal tolerance test.2 Subject will be given breakfast in the form of a mixed meal (10kcal/kg, 45% carbohydrate, 15% protein, 40% fat, 1g/kg glucose) which must be consumed within 15 minutes with glucose, insulin and c-peptide measured from arterialized blood drawn at 0, 10, 20, 30, 60, 90 and 120 minutes from start of meal. From the glucose, insulin and c-peptide measurements calculation of insulin sensitivity (reciprocal of insulin resistance) and β-cell responsivity will be calculated.

Data Collection:

This study will collect demographic information (age, self-described race and ethnicity, sex), and physical data (height, weight, screening blood pressure). Blood and urine samples will be analyzed for various biomarkers to collect the data necessary to carry out the specific aims, as described in the section above. All of these data will be recorded in association with a study identification (ID) number, and kept as secure excel files by the statistician and programmer. The only individually identifiable private data that will be collected are names, addresses, and contact phone numbers so that participants can be screened with follow-up phone calls, and they will be admitted to the inpatient CCI under their name. This personal information, however, will not be associated with the results obtained from the various tests performed, as the latter will be associated with a study ID number. The file linking the study ID number and the personally identifiable information will be kept by the Principal Investigator in a secure location and will not be violated unless it becomes medically necessary to contact a participant on the basis of one of their lab screening tests (e.g., elevated liver function tests).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 30 kg/m2
* Hemoglobin A1c (HbA1c) 6.7-6.4%
* Self reported sleep < 7 hours per night

Exclusion Criteria:

* Inability to extend sleep by one hour each night
* Current or prior history of diabetes OR random serum glucose ≥200mg/dL
* Pregnancy
* Preexisting lung disease requiring oxygen
* Preexisting cardiovascular disease
* Active or uncontrolled psychotic disorder
* Active or uncontrolled bipolar illness
* Active malignancy with in the prior 5 years
* Use of hypoglycemic medication
* estimated glomerular filtration rate (eGFR) <60ml/min/1.73m2
* Use of antihypertensive medications
* Hepatic impairment
* Job requiring rotating overnight shifts
* Bariatric surgery within prior 12 months
* Use of hypnotic medications
* Hematocrit <34% (women), <36% (men)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran J McMullan, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment via posters and online advertisement
Pre-assignment Details: Participants randomization status was not unblinded. All enrolled participants are included in the "melatonin arm"
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 12 | 0
Completed (2 completed visits, however blood samples did not undergo analysis and other measurements were not analyzed.) | 2 | 0
Not Completed | 10 | 0
Not completed — 8 were ineligible | 8 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — PAH not available to study participant | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only two participants completed the trial protocol for reasons detailed elsewhere. Neither of these participants had blood samples or blood pressure measurements analysed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Customized [Count of Participants; unit: Participants]
  Age > 18 years | 12 | 0 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 |  | 8
  Male | 4 |  | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 2 |  | 2
  White | 7 |  | 7
  More than one race | 2 |  | 2
  Unknown or Not Reported | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Renal Specific Renin-aldosterone-angiotensin System (RAAS) Activity
Description: renal specific RAAS activity will be assessed via para-aminohippurate (PAH) renal plasma flow testing with captopril
Time Frame: 6 weeks
Population: Twelve consented participants were screened. Eight were ineligible. One withdrew consent. Only two participants completed the study with blood sampling. One participant was unable to be randomized as PAH was unavailable. For the two participants who completed the study measurements were not made on the samples due to early study termination. The study was terminated due to inability to obtain PAH to perform renal specific RAAS assessments.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Systemic Renin-aldosterone-angiotensin System (RAAS) Activity
Description: systemic RAAS will be assessed by plasma renin activity (PRA), angiotensin II (Ang II) levels and urine aldosterone
Time Frame: 6 weeks
Population: Twelve consented participants were screened. Eight were ineligible. One withdrew consent. Only two participants completed the study. One participant was unable to be randomized as PAH was unavailable. For the two participants who completed the study, measurements were not completed due to early study termination. The study was terminated due to inability to obtain PAH to perform renal specific RAAS assessments.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Glucose Metabolism
Description: Glucose metabolism will be evaluated by applying the Oral Minimal Model method to the results of a 2 hour 7- measurement, mixed meal tolerance test. From the glucose, insulin and c-peptide measurements calculation of insulin sensitivity (reciprocal of insulin resistance) and β-cell responsivity will be calculated.
Time Frame: 6 weeks
Population: Twelve consented participants were screened. Eight were ineligible. One withdrew consent. Only two participants completed the study with blood sampling. One participant was unable to be randomized as PAH was unavailable. For the two participants who completed the study, analysis of measures were not conducted due to early study termination. The study was terminated due to inability to obtain PAH to perform renal specific RAAS assessments.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Central Blood Pressure
Description: Central blood pressure will be measured by pulse wave analysis using the SphygmoCor system (AtCor Medical, West Ryde, NSW, Australia), which measures central blood pressure and arterial stiffness.
Time Frame: 6 weeks
Population: as for outcome 3
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: over 8 weeks
Description: No adverse events were reported
Arm/Group | Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT02631148/Prot_SAP_000.pdf